CLINICAL TRIAL: NCT06974201
Title: An Open Label Study to Determine the Effect of Diabetes M Application Use Versus Conventional Bolus Calculation in Patients With Type 1 Diabetes Mellitus on MDI or CSII
Brief Title: The Effect of Diabetes M Application Use Versus Conventional Bolus Calculation in Patients With Type 1 Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Sofia (Other)
Collaborators: University Hospital for Active Treatment in Endocrinology "Acad Ivan Penchev" EAD (Unknown); Sirma Company (Unknown)
Responsible Party: Principal Investigator, Roumyana Dimova, Assoc Prof, Medical University of Sofia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Approval № 1/2025 MU Sofia
Record Dates: First submitted 2025-04-21; First posted 2025-05-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; bolus calculator
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 30 subjects with type 1 diabetes on MDI or CSII using CGM (Experimental): All subjects enrolled in the trial will be followed-up for 2-weeks on their usual treatment, meaning calculating their bolus insulin doses using conventional bolus calculators and ratios. Then Diabetes M app will be installed and all subjects will be followed-up for 2-weeks using Diabetes M application for calculating their bolus insulin doses.
  Interventions: Device: Diabetes M bolus calculator; Device: Diabetes M app

INTERVENTIONS:
Device: Diabetes M bolus calculator — Diabetes:M Bolus Calculator is an application for precise bolus insulin dose. Full guide for using the Diabetes:M mobile app, can be accessed at
  * In English https://www.manula.com/manuals/sirma-medical-systems/diabetes-m-user- guide/mobile/en/topic/introduction
  * In Bulgarian https://www.manula.com/manuals/sirma-medical-systems/diabetes-m-user- guide/mobile/bg/topic/introduction Instructions for the subject Trial participants must use the Diabetes:M Bolus Calculator before every insulin application and must record the insulin units applied.
  Step-by-step instructions for bolus calculation via Diabetes:M app:
  1. Open Diabetes:M app
  2. Go to Bolus Advisor
  3. Enter blood sugar, carbohydrates
  4. Tap Calculate
  5. Tap Save button
  6. Confirm transferring the bolus to log entry screen
  7. Enter note and some feedback if needed
  8. Tap Save button to save the record
Device: Diabetes M app — Diabetes:M Bolus Calculator is an application for precise bolus insulin dose. Full guide for using the Diabetes:M mobile app, can be accessed at
  * In English https://www.manula.com/manuals/sirma-medical-systems/diabetes-m-user- guide/mobile/en/topic/introduction
  * In Bulgarian https://www.manula.com/manuals/sirma-medical-systems/diabetes-m-user- guide/mobile/bg/topic/introduction Instructions for the subject Trial participants must use the Diabetes:M Bolus Calculator before every insulin application and must record the insulin units applied.
  Step-by-step instructions for bolus calculation via Diabetes:M app:
  1. Open Diabetes:M app
  2. Go to Bolus Advisor
  3. Enter blood sugar, carbohydrates
  4. Tap Calculate
  5. Tap Save button
  6. Confirm transferring the bolus to log entry screen
  7. Enter note and some feedback if needed
  8. Tap Save button to save the record

SUMMARY:
Managing insulin dosing for diabetes, particularly for those with type 1 diabetes mellitus, is a complex process that requires precision. Insulin bolus calculators are designed to help patients calculate their insulin needs based on variables such as carbohydrate intake, blood glucose levels, and insulin sensitivity. However, to ensure these tools are safe and effective, clinical trials are essential. The primary purpose of this trial is to assess the safety and efficacy of the bolus calculator - Diabetes M in providing accurate insulin dosing and preventing the risk of hypoglycemia and hyperglycemia, which can lead to severe complications. The clinical trial is critical to ensure patient's safety and build confidence in the use of the bolus insulin calculator in real-world settings. Insulin dosing errors, whether too high or too low, can lead to serious health risks, including hypoglycemia, hyperglycemia, and long-term diabetes complications. By conducting a controlled study, the trial will evaluate how well the bolus calculator performs in preventing these risks, comparing its recommendations to standard practices. This will help determine whether the calculator can consistently improve blood glucose management while minimizing human error in insulin dosing decisions. Finally, regulatory approval from bodies like the Food and Drug Administration (FDA) requires clear evidence of safety and efficacy. The data from this clinical trial will not only support regulatory submissions but also demonstrate the bolus calculator's clinical utility in improving outcomes like glycemic control and patient compliance. By empowering patients to make more informed dosing decisions and reducing the complexity of diabetes management, this trial could pave the way for broader adoption of this technology and ultimately improve the quality of life for patients with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effect of Diabetes M application use versus conventional bolus calculation (bolus wizard calculation in continuous subcutateous insulin infusion (CSII) or determined insulin:carb ratio (ICR) calculation in multiple daily injections regimen (MDI)) on glycaemic control, measured by time in range (TIR) in percentage defined as time spent in blood glucose levels between 3.9-10.0 mmol/l, in patients with type 1 diabetes on MDI or CSII.

The secondary objectives of this study are: 1) to compare the risk of hypoglycaemic episodes or time below range or time above range (TBR) in percentage, defined as time spent in blood glucose levels between 3.5-3.9 mmol/l level 1 and < 3.5 mmol/l level 2, in patients with type 1 diabetes on MDI or CSII using Diabetes M application versus conventional bolus calculation (bolus wizard calculation in CSII or determined ICR calculation in MDI); 2) to compare the risk of hyperglycaemic episodes or time above range (TAR) in percentage, defined as time spent in blood glucose levels between 10.0-13.0 mmol/l high and >13.0 mmol/l very high, in patients with type 1 diabetes on MDI or CSII using Diabetes M application versus conventional bolus calculation (bolus wizard calculation in CSII or determined ICR calculation in MDI); and 3) to compare time in tight range (TITR) in percentage, defined as time spent in blood glucose levels between 3.9-7.8 mmol/l in patients with type 1 diabetes on MDI or CSII using Diabetes M application versus conventional bolus calculation (bolus wizard calculation in CSII or determined ICR calculation in MDI).

Trial design This is a 4-week, open-label, non-randomized, single-armed, one-centre, proof of concept clinical trial. All subjects enrolled in the trial will be followed-up for 2-weeks on their usual treatment and then Diabetes M app will be applied. There is a 2-week screening period followed by enrolment visit (V1). At V1 venuos blood samples will be taken for laboratory tests all participants from all participants. Then there is a 2-week follow-up period on usual treatment ending with visit 2 (V2) when CGM data for the period will be downloaded and Diabetes M application will be installed. All individual parameters for the participants will be filled in the application and the participants will be instructed in details on how to use the application. Then there is a 2-week treatment period using Diabetes M application ending with visit 3 (V3) when CGM data for the period will be downloaded. Total trial duration for the individual subject will be approximately 6 weeks. The trial population will consist of subjects with type 1 diabetes treating with MDI or CSII and using continuous glucose monitoring (CGM).

Subject and trial completion Approximately 40 subjects will be screened in order to achieve 30 subjects to be assigned. The number of subjects expected to complete the trial will be 27 subjects (calculated 10% drop-off). Subjects will be followed for the planned duration of the trial.

Trial period completion for a subject is defined as when the enrolled subject has completed the final scheduled visit 'end of trial', visit 3. Date of trial completion is the date the subject completed the final scheduled visit, as mentioned above.

Treatment period completion for a subject is defined as when the subject has received the required treatment and attended the end of treatment visit 3.

Scientific rationale for trial design The treatment duration of the trial is 4 weeks, including 2 weeks on conventional bolus calculation and 2 weeks on Diabetes M app. A 2-week treatment duration is comparable to trials conducted with a previously approved device, which will serve as a predicator in the current study, and will provide robust data for the evaluation of efficacy and safety parameters. This open-label, non-randomized, single-armed, one-centre, proof of concept clinical trial design has the poor to accurately assess the effect and safety of Diabetes M application as an alternative bolus calculator in subjects with type 1 diabetes on MDI or CSII. The trial includes a screening visit to assess the subject's eligibility. After enrollment visit, there are 2 visits scheduled. Visit 2 is scheduled 2 weeks after enrolment for switching from conventional treatment to Diabetes M app installation and use. An end of trial visit 3 for efficacy and safety assessments is scheduled 2 weeks after visit 2.

The trial population will consist of subjects with type 1 diabetes on treatment with MDI or CSII using CGM. Patients with type 1 diabetes represent a clinically relevant high-risk population and it is highly likely to benefit from the use of such an application.

Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, is not permitted.

Full guide for using the Diabetes:M mobile app, can be accessed at

* In English https://www.manula.com/manuals/sirma-medical-systems/diabetes-m-user- guide/mobile/en/topic/introduction
* In Bulgarian https://www.manula.com/manuals/sirma-medical-systems/diabetes-m-user- guide/mobile/bg/topic/introduction Auxiliary supplies

The following auxiliary supplies will be provided by investigators:

* Glucometer and blood strips for calibration if needed
* Three refills of CGM sensors Dexcom One plus (each lasts 10 days for a total of 30 days or 4 weeks). The study requires that participants use the standard Dexcom mobile app and that the Primary Investigator can download their daily data from the physician online access provided by Dexcom.

Only supplies provided by investigators must be used for the administration of the trial product.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to be included in the trial only if all the following criteria apply:

  1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
  2. Ability to adhere to the study visit schedule and other protocol requirements.
  3. Male or female, age from 18 years to 75 years at the time of signing informed consent.
  4. Diagnosed with type 1 diabetes regardless of the disease duration.
  5. On treatment with MDI or CSII.
  6. Using CGM.
  7. eGFR-EPI ≥ 45 ml/min/1.73m 2 .

Exclusion Criteria:

* Subjects are excluded from the trial if any of the following criteria apply:

Diabetes related

1. Male or female, age < 18 years or > 75 years. 2. Diagnosed with type 2 diabetes. 3. Diagnosed with diabetes proliferative retinopathy. 4. Renal impairment measured as estimated glomerular filtration rate (eGFR-EPI) value of < 45 mL/min/1.73 m 2 according to KDIGO. 5. Frequent severe hypoglycaemic episodes (<3.5 mmol/l). 6. Any acute illnesses, which might influence glycaemic control in short term. General safety 8. Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 3 months prior to the day of screening. 9. Presently classified as being in New York Heart Association (NYHA) Class IV. 10. Presence or history of malignant neoplasm within 5 years prior to the day of screening.

11. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method. 12. Any disorder, unwillingness or inability, which in the investigator's opinion, might jeopardise the subject's safety or compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Change from first phase (week 0-2) to second phase (week 3-4) in TIR (%) | From enrollment to the end of treatment at 4 weeks.
  The primary outcome measure is defined as a change in time in range (3.9-10 mmol/l) for glucose between the two estimated periods: the first period without using Diabetes M application for bolus insulin calculation and the second period with using Diabetes M application for bolus insulin calculation.

SECONDARY OUTCOMES:
Change from first phase (week 0-2) to second phase (week 3-4) in TBR (%) | From enrollment to the end of treatment at 4 weeks.
  The secondary outcome measure is defined as a change in time below range (<3.9 mmol/l) for glucose between the two estimated periods: the first period without using Diabetes M application for bolus insulin calculation and the second period with using Diabetes M application for bolus insulin calculation.
Change from first phase (week 0-2) to second phase (week 3-4) in TAR (%) | From enrollment to the end of treatment at 4 weeks.
  The secondary outcome measure is defined as a change in time above range (>10.0 mmol/l) for glucose between the two estimated periods: the first period without using Diabetes M application for bolus insulin calculation and the second period with using Diabetes M application for bolus insulin calculation.
Change from first phase (week 0-2) to second phase (week 3-4) in TITR (%) | From enrollment to the end of treatment at 4 weeks.
  The secondary outcome measure is defined as a change in time in tight range (3.9-7.8 mmol/l) for glucose between the two estimated periods: the first period without using Diabetes M application for bolus insulin calculation and the second period with using Diabetes M application for bolus insulin calculation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital for Active Treatmnet in Endocrinology "Acad Ivan Penchev" EAD, Medical University of Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No